CLINICAL TRIAL: NCT02993432
Title: High Volume Foleys Increasing Vaginal Birth (High FIVe Birth) Pilot Trial
Brief Title: High Volume Foleys Increasing Vaginal Birth Pilot Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: AFP Innovation Fund (Other)
Responsible Party: Principal Investigator, Dr. Anne Berndl, Assistant Professor University of Toronto Division of Maternal Fetal Medicine Department of Obstetrics and Gynaecology, Associate Scientist, Sunnybrook Research Institute, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SHS-16-002
Record Dates: First submitted 2016-12-05; First posted 2016-12-15 (Estimated); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Labour; Induced; Pilot Study; Cervical Ripening
MeSH Terms: interventions — KLK15 protein, human; Dinoprostone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prostaglandin (Active Comparator): Administration of the prostaglandin for cervical ripening of the clinician's choice, ie Prostin (Prostin E2 Vaginal Gel 1mg intravaginally) or Cervidil (dinoprostone, 10 mg vaginal insert)
  Interventions: Drug: prostaglandin of the clinician's choice
- Foley catheter filled to 80cc (Experimental): Insertion of a Foley catheter through the cervix and filling to 80cc
  Interventions: Device: Foley catheter filled to 80cc

INTERVENTIONS:
Device: Foley catheter filled to 80cc — A Foley catheter is inserted through the cervix and filled to 80cc
  Arms: Foley catheter filled to 80cc
Drug: prostaglandin of the clinician's choice — Insertion of the prostaglandin (Prostin (1mg dinoprostone vaginal gel) or Cervidil (10mg vaginal slow release insert)) of the clinicians choice into the vagina for the purpose of cervical ripening
  Other Names: Prostin, Cervidil
  Arms: Prostaglandin

SUMMARY:
It is currently unknown if there is a way to decrease the risk of cesarean delivery when undergoing cervical ripening and induction of labour. Some research suggests a Foley catheter placed through the cervix and filled to 80cc may decrease this risk. We wish to run a large scale trial to see if Foleys filled to 80cc decrease the risk of Cesarean section compared to the commonly used medication for cervical ripening, prostaglandins. Before we can undertake a large trial, we need to do a pilot to see if women will agree to participate in this type of study. As well, a pilot will help with trouble shooting prior to a large trail, to improve the chances of successfully answering this clinically important question.

DETAILED DESCRIPTION:
Background:

Approximately 1/3 of first-time mothers (nulliparous women) undergoing induction of labour deliver by cesarean. Cesarean delivery can have negative consequences to the initial and subsequent pregnancies. Women who have a cesarean in their first pregnancy are more likely to have a cesarean in their following pregnancies and this group is the largest contributor to the overall cesarean delivery rate. Therefore, targeting interventions that prevent cesareans in nulliparous women undergoing induction of labour will have a substantial impact on the overall cesarean delivery rate.

Adequate ripening or preparing the cervix before induction has been found to decrease the risk of cesarean. This can be done by a variety of methods, such as prostaglandins (a chemical messenger) or a Foley filled to a moderate volume of fluid. These methods have been found to be equal regarding the risk of cesarean delivery. However, a meta-analysis by our team discovered a trend towards a decreased risk of cesarean when cervical ripening is undertaken with Foleys filled to a high volume of fluid (80cc) compared to those filled to a low volume (30cc).Most Canadian Obstetricians use prostaglandins for cervical ripening. To assess if 80cc Foleys result in a lower risk of cesarean, they need to be compared to the Canadian standard of prostaglandins. Therefore a randomized controlled trial is required.

The Greater-Toronto-Area Obstetric (GTA-OB) Network is a group of hospitals committed to facilitating research and will be the setting for the planned large scale trial. The large scale trial will aim to demonstrate a difference in the rate of cesarean from 38% to 31%, which will require the enrollment of 1442 women. It has been estimated that there are 5,437 women who will meet entry criteria in the GTA-OB network each year, if ½ are approached, 20% will need to consent to complete the trial in 3 years. Therefore, this pilot study will determine if this recruitment rate is potentially achievable and will inform design strategies to ensure its success.

The discovery of a simple, non- pharmacological, cost effective manner of cervical ripening that decreases the risk of cesarean would change clinical practice and significantly improve safety for the 33,000 Canadian women and their babies who undergo cervical ripening each year. This pilot trial is a crucial step towards this discovery.

Objectives:

The primary objective for this pilot trial is to determine the probability that an eligible woman will agree to be randomized into the trial comparing 80cc Foleys to prostaglandins for cervical ripening. This study aims to assess if it is possible to obtain a recruitment rate of 20%.

The secondary objective will be a systematic evaluation of the pilot trial process to guide full-scale study design.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous women 37 weeks and 0 days to 41 weeks and 6 days gestational age (term) requiring cervical ripening
* Health care provider feels it is possible to administer either method of cervical ripening.
* Bishop score of 6 or less
* Live, singleton, cephalic fetus
* Availability of personnel to consent and randomize participants

Exclusion Criteria:

* Non-viable fetus
* Contraindication to cervical ripening, labour induction or labour
* Prior attempt at induction of labour in this pregnancy
* Spontaneous rupture of fetal membranes
* Evidence of labour or regular uterine contractions
* Lack of consent

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2016-12; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
The percentage of eligible women who are approached to participate in the study that are enrolled and randomized to either the use of a high volume Foley or prostaglandin for cervical ripening | 15 months
  The primary outcome measure of percent of women recruited will be captured by the number of women who undergo the randomized intervention divided by the number of women who are approached.

CONTACTS AND LOCATIONS:
Overall Officials: Anne ML Berndl, MD MSc, Principal Investigator — Sunnybrook Health Sciences Centre,University of Toronto

IPD SHARING:
Plan to Share IPD: No
There is not currently an IPD sharing plan

REFERENCES:
- [Background] Berndl A, El-Chaar D, Murphy K, McDonald S. Does cervical ripening at term using a high volume foley catheter result in a lower caesarean section rate than a low volume foley catheter? A systematic review and meta-analysis. J Obstet Gynaecol Can. 2014 Aug;36(8):678-687. doi: 10.1016/S1701-2163(15)30509-0. PMID 25222162
- [Background] Leduc D, Biringer A, Lee L, Dy J; CLINICAL PRACTICE OBSTETRICS COMMITTEE; SPECIAL CONTRIBUTORS. Induction of labour. J Obstet Gynaecol Can. 2013 Sep;35(9):840-857. doi: 10.1016/S1701-2163(15)30842-2. English, French. PMID 24099451
- [Background] Jozwiak M, Bloemenkamp KW, Kelly AJ, Mol BW, Irion O, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2012 Mar 14;(3):CD001233. doi: 10.1002/14651858.CD001233.pub2. PMID 22419277
- [Background] Levy R, Kanengiser B, Furman B, Ben Arie A, Brown D, Hagay ZJ. A randomized trial comparing a 30-mL and an 80-mL Foley catheter balloon for preinduction cervical ripening. Am J Obstet Gynecol. 2004 Nov;191(5):1632-6. doi: 10.1016/j.ajog.2004.03.033. PMID 15547534
- [Background] Kashanian M, Nazemi M, Malakzadegan A. Comparison of 30-mL and 80-mL Foley catheter balloons and oxytocin for preinduction cervical ripening. Int J Gynaecol Obstet. 2009 May;105(2):174-5. doi: 10.1016/j.ijgo.2009.01.005. Epub 2009 Feb 20. No abstract available. PMID 19232606
- [Background] Delaney S, Shaffer BL, Cheng YW, Vargas J, Sparks TN, Paul K, Caughey AB. Labor induction with a Foley balloon inflated to 30 mL compared with 60 mL: a randomized controlled trial. Obstet Gynecol. 2010 Jun;115(6):1239-1245. doi: 10.1097/AOG.0b013e3181dec6d0. PMID 20502296
- [Background] Jozwiak M, Oude Rengerink K, Benthem M, van Beek E, Dijksterhuis MG, de Graaf IM, van Huizen ME, Oudijk MA, Papatsonis DN, Perquin DA, Porath M, van der Post JA, Rijnders RJ, Scheepers HC, Spaanderman ME, van Pampus MG, de Leeuw JW, Mol BW, Bloemenkamp KW; PROBAAT Study Group. Foley catheter versus vaginal prostaglandin E2 gel for induction of labour at term (PROBAAT trial): an open-label, randomised controlled trial. Lancet. 2011 Dec 17;378(9809):2095-103. doi: 10.1016/S0140-6736(11)61484-0. Epub 2011 Oct 24. PMID 22030144
- [Derived] de Vaan MD, Ten Eikelder ML, Jozwiak M, Palmer KR, Davies-Tuck M, Bloemenkamp KW, Mol BWJ, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD001233. doi: 10.1002/14651858.CD001233.pub4. PMID 36996264

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-22): https://cdn.clinicaltrials.gov/large-docs/32/NCT02993432/Prot_SAP_000.pdf